CLINICAL TRIAL: NCT01401777
Title: Electromagnetic Tracking of Devices During Interventional Procedures - A Cryoablation Study
Status: Withdrawn | Type: Observational
Why Stopped: On hold pending product development
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010_CRYO_V7
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Kidney Tumors
Keywords: Kidney Tumors, Cryoablation, Biopsy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control, No PercuNav: Patient having procedure without PercuNav Guidance information
- PercuNav aided procedure: Biopsy procedure aided with use of PercuNav

SUMMARY:
The objective of this study is to assess and quantify any differences between assisted (using real-time visualization of tracked cryo-probes) and unassisted cryoablation procedures using pre-procedure CT scans or CT fluoroscopy with respect to:

Primary Endpoint:

• "TRE" Target Registration Error (distance between "virtual" needle position (tracking data) and the actual needle position (CT confirmation scan))

Secondary Endpoints

* Accuracy of needle targeting - The vector of each needle insertion (The initial vector allows us to project the path to the pre-defined target. If the initial entry point is not ideal, the path to the target will need adjustment) Based on a two-sample t-test (significance level of 0.05, two-tailed), the study has 89% power to detect a difference of 2mm in accuracy between the two treatment groups (assuming a standard deviation of 1.9mm).
* Measure time difference between assisted and unassisted procedure

DETAILED DESCRIPTION:
The objective of this study is to assess and quantify any differences between assisted (using real-time visualization of tracked cryo-probes) and unassisted cryoablation procedures using pre-procedure CT scans or CT fluoroscopy. To assess this, physicians will perform ablation procedures with and without the Percu Nav device. Data will be collected on the angle of needle entry unassisted and then assisted by PercuNAv to determine if the added imaging information modifies the physician's needle approach.

Each patient will have a pre-procedure CT image set of the area of interest acquired. The patient will be scanned in the same position that the ablation will be performed in, although not requisite. Sterile registration patches will be applied to the patient's skin around the area of interest prior to the scan, ensuring that suitable windows are left available for needle entry. The patient will undergo these pre-procedural scans as part of the usual clinical evaluation of the lesion to undergo ablation. The scans may be acquired with or without contrast, at the discretion of the physician.

Control group: The physician will perform the procedure using the standard of care method (CT only), without the additional information being recorded by the PercuNav device. The tracking device will be placed on the patient's skin at the desired point of entry. Without displaying the PercuNav screen to the physician, a screen capture will be taken to record the approach path. At the point of insertion, the time stamp will be recorded and the start button will be pressed. Once the physician states they are at the defined target a screen capture will be taken on the PercuNav and the distance to target and time stamp will be recorded by pushing the start button again. At the end of the procedure a verification CT scan will be taken with the needle in place and sent to the PercuNav.

Percu Nav group: The physician will perform the procedure using the standard of care procedure with the additional information displayed and recorded by the PercuNav device (CT and PercuNav). The tracking device will be placed on the patient's skin at the desired point of entry. Without displaying the PercuNav screen to the physician, a screen capture will be taken to record the approach path. The physician will be shown the PercuNav screen and will correct the desired approach path and another screen capture will be taken. At the point of insertion, the time stamp will be recorded and the start button will be pressed. Once the physician states they are at the defined target a screen capture will be taken on the PercuNav and the distance to target and time stamp will be recorded. At the end of the procedure a verification CT scan will be taken (as is part of the regular standard of care procedure) with the needle in place and sent to the PercuNav.

The outcome measures that will be evaluated in the groups include:

1. Accuracy - The distance between the "virtual" needle position (tracking data) and the actual needle position (CT confirmation scan)), where applicable (TRE)
2. Time to reach a clinically acceptable target in the tumor
3. The total procedure time
4. Accuracy of needle targeting - The vector of each needle insertion (The initial vector allows us to project the path to the pre-defined target. If the initial entry point is not ideal, the path to the target will need adjustment)

ELIGIBILITY:
Inclusion Criteria:

1. Has had a pre-operative CT/MRI scan performed and will be undergoing an ablation procedure of the kidney;
2. Is over the age of 18;
3. Has the ability to understand and the willingness to sign a written informed consent form, and complies with the protocol;
4. Has the ability to follow procedural instructions, including, but not limited to, holding their breath and remaining reasonably motionless during the procedure.

Exclusion Criteria:

1. Was precluded from an ablation procedure based on standard ablation exclusions; 2. Has an adhesive allergy (due to the application of active fiducials with adhesive backing); 3. Has a pacemaker or automatic implantable cardiac defibrillator; 4. Has a gross body weight above the procedural table limit (typically > 170 kg); 5. Is pregnant

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Promary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Target Registration Error | 24 hrs
  "TRE" Target Registration Error (distance between "virtual" needle position (tracking data) and the actual needle position (CT confirmation scan))

SECONDARY OUTCOMES:
Accuracy of needle targeting | 24 hrs
  The vector of each needle insertion (The initial vector allows us to project the path to the pre-defined target. If the initial entry point is not ideal, the path to the target will need adjustment)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States